CLINICAL TRIAL: NCT04413175
Title: A Randomized Controlled Trial on the Effects of Music Therapy on Procedural Pain, Anxiety and Comfort Level During Cystoscopy
Brief Title: Effects of Music Therapy on Procedural Pain, Anxiety and Comfort Level During Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hanife DURGUN, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HanifeD
Record Dates: First submitted 2020-05-18; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Cystoscopy
Keywords: Anxiety; comfort; cystoscopy; music therapy; pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a music group (Experimental): Patients in the music group were provided music therapy that was prepared by the Turkish Psychological Association. They listened to the music that has a calming and relaxing effect for 20 min before and during the procedure.
  Interventions: Other: music therapy
- control group (No Intervention): control group

INTERVENTIONS:
Other: music therapy — Patients in the music group were provided music therapy that was prepared by the Turkish Psychological Association. They listened to the music that has a calming and relaxing effect for 20 min before and during the procedure.
  A portable MP3 player connected to double earphones was used in the present study. After patients took the lithotomy position for cystoscopy, their headphones were inserted and music began to be played. Music was played to the individuals for 20 minutes before and during the procedure. Headphones were removed immediately after the procedure was completed and the double earphones were cleaned with antiseptic solution after each application.
  Arms: a music group

SUMMARY:
Aims and objectives: This study aimed to determine the effect of music therapy on procedural pain intensity and anxiety and comfort levels in patients during cystoscopy.

Background: Cystoscopy is a procedure that is commonly performed as day surgery in urology clinics in order to diagnose lower urinary tract system symptoms as well as to diagnose and follow up tumors associated with the lower urinary system. During cystoscopy, which is an invasive intervention, individuals may experience pain and anxiety, and their comfort may be negatively affected.

Methods: This study was a prospective, randomized controlled trial. Study participants were randomly assigned to either a control or music group. The outcome measures were assessed using the Visual Analogue Scale, State Anxiety Scale, and General Comfort Questionnaire. This report followed the CONSORT checklist.

DETAILED DESCRIPTION:
1. INTRODUCTION Cystoscopy is a common procedure in urology clinics and has two types: flexible and rigid. Especially recently, there has been an increase in the use of flexibles. Both of these types can be preferred as a diagnostic procedure in hematuria, atypical dysuria, bladder and upper urinary tract cancers, and suspected urethral stenosis. Rigid cystoscopy can be more painful than flexible cystoscopy.
2. BACKGROUND Cystoscopy is a procedure performed in urology clinics to evaluate the lower urinary tract for a large number of symptoms and pathologies, but it is painful and causes anxiety in individuals. It is recommended to perform local anesthesia to the patients during the procedure, to select appropriate cystoscopy equipment, and to make the necessary environmental arrangements in order to reduce the patients' pain and anxiety and increase their comfort levels.

Environmental arrangements to manage interventional pain in cystoscopy include music therapy that has recently been used widely.Music is used as one of the complementary therapies in the treatment of many diseases due to its physical, psychological, and functional effects on individuals. The use of music as therapy in hospitals began to become widespread with the beginning of the world wars, but the introduction of pharmacological methods for the treatment of pain and anxiety has reduced the popularity of music in this context. With the identification of side effects of drugs in the subsequent years, starting again to use music as complementary therapy has come to the fore.

Music therapy in nursing first started in the 1800s with Florence Nightingale. Nightingale described music as an effective method in the recovery process in order to provide and increase patient comfort and reduce their anxiety levels. Music therapy has also been accepted as part of nursing practices within the scope of Nursing Interventions Classification.

In the literature, international studies have been conducted to reduce the pain and anxiety levels of individuals and increase their comfort levels. Considering two systematic reviews related to the subject;some studies noted that music played during flexible cystoscopy did not reduce pain and anxiety, while some studies stated that music could be effective in reducing pain and anxiety during cystoscopy. Controversial results were found in these two studies, which have high evidence levels. Experimental studies with control groups showed that music reduced pain and anxiety and increased comfort levels in patients undergoing flexible cystoscopy. Given the limitations of the studies on the subject and sample power/deficiencies, it may be observed that controversial conclusions have been reached about the effectiveness of music in relieving pain and anxiety. On the other hand, only one study has been found in Turkey regarding this issue. In a study, the effects of various distraction methods applied during the cystoscopy procedure (group 1: music, group 2: stress ball, group 3: video, and group 4: control) on pain, anxiety, and satisfaction were examined. The study found that the patients in the video group had lower pain and anxiety levels than those in the other groups. Considering the national and international studies available in the literature, regarding the topic of music therapy that may be effective in reducing pain and anxiety during the cystoscopy procedure, it is necessary to conduct further studies that provide high levels of evidence and produce scientific knowledge with greater sample sizes and by using randomized-controlled trials that are fundamental in assessing the effectiveness of evidence-based practices. This study aimed to determine the effect of music therapy on procedural pain intensity and anxiety and comfort levels in patients during cystoscopy.

2.1. Study hypotheses Hypothesis 1. Music therapy reduces procedural pain in patients during cystoscopy.

Hypothesis 2. Music therapy reduces anxiety in patients during cystoscopy. Hypothesis 3. Music therapy increases comfort level in patients during cystoscopy.

ELIGIBILITY:
Inclusion criteria:

* Patients older than 18 years,
* Being literate,
* Having no hearing problems.

Exclusion criteria:

* Patients who had allergies to anesthetic drugs
* Urinary tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Pain scores | before cystoscopy
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain scores | during cystoscopy procedure
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Pain scores | immediately after cystoscopy procedure is completed
  The primary outcome of the study was to measure pain using a 10-cm VAS, with high numbers meaning greater pain intensity. The VAS is used to measure various subjective clinical phenomena, including pain. It is quick and easy to use and score. The 0-10 VAS requires the patients to choose a number from 0 to 10 that best represents their pain; 0 is the equivalent of "no pain," and 10 is the equivalent of the worst imaginable pain
Anxiety score | before cystoscopy
  Anxiety was used as the secondary outcome and measured using the Turkish version of the State-Trait Anxiety Inventory (STAI). The inventory was developed by Spielberger and colleagues and tested for its validity and reliability in Turkish by Öner and Le Compte. Its internal consistency, test-retest reliability, and item-by-item reliability values were found to be between 0.83 and 0.87, 0.71 and 0.86, and 0.34 and 0.72, respectively. The STAI consists of a State Anxiety Scale (STAI-S) and a Trait Anxiety Scale (STAI-T). Only the STAI-S was used in this study. The lowest total score that can be obtained from the scale is 20, and the highest total score is 80. A high score indicates high anxiety level, and a low score indicates low anxiety level
Anxiety score | immediately after cystoscopy procedure is completed
  Anxiety was used as the secondary outcome and measured using the Turkish version of the State-Trait Anxiety Inventory (STAI). The inventory was developed by Spielberger and colleagues and tested for its validity and reliability in Turkish by Öner and Le Compte. Its internal consistency, test-retest reliability, and item-by-item reliability values were found to be between 0.83 and 0.87, 0.71 and 0.86, and 0.34 and 0.72, respectively. The STAI consists of a State Anxiety Scale (STAI-S) and a Trait Anxiety Scale (STAI-T). Only the STAI-S was used in this study. The lowest total score that can be obtained from the scale is 20, and the highest total score is 80. A high score indicates high anxiety level, and a low score indicates low anxiety level
Comfort scores | before cystoscopy
  The third outcome was comfort, which was measured using the General Comfort Questionnaire (GCQ). This questionnaire was developed by Katharine Kolcaba to determine individuals' comfort needs and evaluate nursing interventions that may be employed to ensure and increase such comfort. The GCQ uses a four-point Likert-type scale and consists of 48 items. The lowest score that can be obtained when using the scale is 48, and the highest score is 192. The GCQ was adapted for use in a Turkish context by Kuğuoğlu and Karabacak.
Comfort scores | immediately after cystoscopy procedure is completed
  The third outcome was comfort, which was measured using the General Comfort Questionnaire (GCQ). This questionnaire was developed by Katharine Kolcaba to determine individuals' comfort needs and evaluate nursing interventions that may be employed to ensure and increase such comfort. The GCQ uses a four-point Likert-type scale and consists of 48 items. The lowest score that can be obtained when using the scale is 48, and the highest score is 192. The GCQ was adapted for use in a Turkish context by Kuğuoğlu and Karabacak.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Durgun, Dr, Principal Investigator — Ordu State Hospital
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No